CLINICAL TRIAL: NCT05138939
Title: Effects of Japanese Red Wines on Vascular Function in Adult Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1306528
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Vascular Function; Platelet Aggregation
Keywords: vascular function; platelet aggregation

STUDY DESIGN:
Intervention Model Description: Three-way crossover randomized controlled trial
Who Masked: Participant
Masking Description: Participants will be blinded by the type of beverages (control, red wine1, and red wine2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Participants in this group are randomized to receive Isocaloric beverage (a beverage that has similar caloric content to the red wines) as the first intervention.
  Interventions: Other: Red wine A; Other: Red wine B; Other: Control
- Red wine A (Experimental): Participants in this group are randomized to receive red wine A as the first intervention (can be the younger or older vintage).
  Interventions: Other: Red wine A; Other: Red wine B; Other: Control
- Red wine B (Experimental): Participants in this group are randomized to receive red wine B as the first intervention (can be the younger or older vintage)
  Interventions: Other: Red wine A; Other: Red wine B; Other: Control

INTERVENTIONS:
Other: Red wine A — 8 oz (237 ml) of red wine A and red wine B will be blinded and randomized between Japanese Zweigelt red wines from vintages 2015 or 2018.
Other: Red wine B — 8 oz (237 ml) of red wine A and red wine B will be blinded and randomized between Japanese Zweigelt red wines from vintages 2015 or 2018.
Other: Control — 8 oz (237 ml) of control beverage is a beverage that has similar calories to red wines.

SUMMARY:
The overall objective of this study is to investigate the effects of different types of red wine on markers of endothelial function and platelet aggregation.

DETAILED DESCRIPTION:
Potential participants are provided with information about the study and potential risks. Once participants decided to participate in the study, they will be scheduled for a health screening visit which determines eligibility to the study entry. If participants are eligible, they will be randomized in a three-way crossover study design to receive three interventions (control, red wine1, and red wine2) with the one-week washout period. On the study day, participants will be assessed for baseline measurements, provided with the designated beverage, and followed up for the measurements at 2 and 4 hours after the consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male: 50-70 years old
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* BMI 18.5 - 40 kg/m2
* Weight ≥ 110 pounds
* Prescription medication if on a 6-month self-reported stable dose
* Regularly consume alcoholic beverages (2 drinks/week to 2 drinks/day)
* Non-smokers
* One standard drink of alcoholic beverages is defined as follow:

  12-ounces of beer (5% alcohol content) (~1 regular bottle). 8-ounces of malt liquor (7% alcohol content) (~1 regular bottle). 5-ounces of wine (12% alcohol content) (~½ glass) 1.5-ounces of 80-proof (40% alcohol content) distilled spirits or liquor (e.g., gin, rum, vodka, whiskey) (~ 1 shot)

Exclusion Criteria:

* BMI ≥ 40 kg/m2
* Daily use of aspirin or NSAIDs
* Dislike or allergic to any food, especially wine, grape, and alcohol
* Vegan, Vegetarians, food faddists, or those consuming a non-traditional diet
* Alcohol consumption < 2 drinks/week (i.e. 1 bottle of beer, ½ glass of wine, and 1 shot of hard liquor)
* Alcohol consumption > 2 drinks/ day
* Fruit consumption ≥ 2 cups/day
* Vegetable consumption ≥ 3 cups/day
* Fatty Fish ≥ 3 times/week
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and Stroke
* Self-reported Cushing's syndrome
* Self-reported chronic/routine high-intensity exercise
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Liver or Chemistry panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within the past 5 years
* Self-reported malabsorption
* Use of multi-vitamin and minerals other than a general formula of vitamins and minerals that meet the recommended dietary allowance (RDA)
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Current enrollee in a clinical research study.
* Reactive hyperemia index (RHI) value ≥ 2.8 (measured by PAT at the first study visit)
* Raynaud's disease, history of bleeding disorder and/or abnormal bleeding, and history of gastrointestinal ulceration and/or bleeding
* Under current medical supervision
* 1 ug/ml and 3 ug/ml collagen screening maximal platelet aggregatory response of < 65%.
* Platelet number or mean platelet values that are outside of the normal reference range as indicated on a complete blood cell count report from the University of California Davis Medical Center
* Current diagnosis of anemia; or a screening hemoglobin and hematocrit that is less than the normal reference range.Individuals with blood clotting or platelet defect disorders

The following special populations will be excluded:

* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-02-04 (Actual); Study Completion 2023-02-04 (Actual)

PRIMARY OUTCOMES:
Peripheral Arterial Tonometry (PAT) | Baseline
  Endothelial function
Peripheral Arterial Tonometry (PAT) | 2 hours after beverage consumption
  Endothelial function
Peripheral Arterial Tonometry (PAT) | 4 hours after beverage consumption
  Endothelial function

SECONDARY OUTCOMES:
Platelet Aggregation | Baseline and 2 and 4 hours after beverage consumption
  Light Transmission Aggregometry

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Hackman, PhD, Principal Investigator — Department of Nutrition, UC Davis
Locations (1):
- Ragle Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No